CLINICAL TRIAL: NCT06081673
Title: A Phase II Clinical Study of Penpulimab Combined With Chemotherapy for Neoadjuvant and Adjuvant Therapy in Patients With Resectable Head and Neck Squamous Cell Carcinoma
Brief Title: Penpulimab Combined With Chemotherapy for Neoadjuvant and Adjuvant Therapy in Patients With Resectable HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-HN001
Record Dates: First submitted 2023-09-25; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — penpulimab; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penpulimab combined with cisplatin and albumin-paclitaxel neoadjuvant therapy (Experimental): Penpulimab injection combined with cis-platinum and albumin-bound paclitaxel before surgery, 21 days as a treatment cycle.
  Adjuvant therapy was started within 6 weeks after surgery：Patients who achieved MPR after surgery were randomized 1:1 with standard adjuvant therapy(RT alone or combined with cisplatin) and Alternative adjuvant therapy(RT alone or combined with Penpulimab).
  Non-MPR patients receive standard adjuvant therapy
  Interventions: Drug: Penpulimab injection; Drug: cisplatin; Drug: albumin-paclitaxel

INTERVENTIONS:
Drug: Penpulimab injection — Penpulimab is a human immunoglobulin G1(IgG1) monoclonal antibody (mAb) directly programmed cell death-1 (PD-1). AK105 can effectively prevent human PD-1 binds to programmed cell death-1 ligand 1(PD-L1) and programmed cell death-1 ligand 2(PD-L2)； 200mg,D1, IV(21 days/cycle).
Drug: cisplatin — Cisplatin :75mg/m2, D1, IV(21 days/cycle)
Drug: albumin-paclitaxel — albumin-paclitaxel :260mg/m2,IVgtt,D1(21 days/cycle)

SUMMARY:
This study aims to observe and explore the efficacy and safety of Penpulimab combined with chemotherapy for neoadjuvant and adjuvant therapy in patients with resectable head and neck squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily joined the study, signed the informed consent, and had good compliance;
* Patients with 18 Years to 75 Years(at the time of signing the informed consent); Eastern Cooperative Oncology Group Performance Status (ECOG-PS) score: 0-1;
* Patients with untreated head and neck squamous cell carcinoma who were pathologically confirmed and determined to be suitable for surgical treatment were classified as stage III, IVa according to AJCC (8th Edition), including oral, oropharyngeal, hypopharyngeal, and laryngeal cancers
* Female patients of reproductive age should agree that birth control (such as intrauterine device, birth control pills, or condoms) must be used during the study period and for six months after completion; Having a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating; Male patients should agree to use contraception during the study period and for six months after the end of the study.

Exclusion Criteria:

* Patients who have previously used PD-1/PD-L1/CTLA-4 antibody therapy;
* Patients who require systemic treatment with corticosteroids (> 10mg daily prednisone equivalent) or other immunosuppressive drugs within 14 days prior to administration or during treatmentIn the absence of active autoimmune disease, inhaled or topical steroids and adrenocortical hormone at doses >10mg/ day equivalent to prednisone and adrenocortical hormone replacement at therapeutic doses not exceeding 10mg/ day prednisone are permitted;
* A history of any active immune or autoimmune disease, or a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Active or uncontrolled severe infection within 4 weeks prior to enrollment (CTCAE grade 2 infection);
* Abnormal function of major organs
* Patients with concomitant diseases that, in the investigator's judgment, may seriously endanger patients' safety or may interfere with the completion of the study, or are deemed unsuitable for inclusion for other reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-10-30 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Major pathological response（MPR） | One year
  Major pathologic response is based on the pathological examination on the post-operative specimens.

SECONDARY OUTCOMES:
Disease-control Rate（DCR） | Baseline up to 3 years.
  The proportion of subjects response of CR, PR, or SD (subjects achieving SD will be included in the DCR if they maintain SD for ≥4 weeks).
Adverse event rate | Baseline up to 3 years.
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Disease-free survival at 2 years(DFS at 2 years) | Baseline up to 2 years.
  The proportion of subjects disease-free survival at 2 years
Overall Response Rate (ORR) | Baseline up to 3 years.
  The proportion of subjects who achieves a best overall response of CR or PR.
Local recurrence-free survival at 2years(LRFS at 2 years) | Baseline up to 2 years.
  The proportion of subjects local recurrence-free survival at 2years
distant metastasis-free survival at 2 years(DMFS at 2 years) | Baseline up to 2 years.
  The proportion of subjects distant metastasis-free survival at 2years
OS at 2 years | Baseline up to 2 years.
  The overall survival time refers to the time from initiating inductive therapy to death due to any cause.
pathologic complete response(pCR) | One year
  Pathological examination showed the presence of 0% active tumor in the tissue specimen

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hostipal, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China